CLINICAL TRIAL: NCT02729051
Title: A Phase IIIB, 24-week Randomised, Double-blind Study to Compare 'Closed' Triple Therapy (FF/UMEC/VI) With 'Open' Triple Therapy (FF/VI + UMEC), in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Comparative Study of Fluticasone Furoate(FF)/Umeclidinium Bromide (UMEC)/ Vilanterol (VI) Closed Therapy Versus FF/VI Plus UMEC Open Therapy in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200812; 2015-005212-14 (EudraCT Number)
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD); fluticasone furoate/umeclidinium bromide/vilanterol (FF/UMEC/VI); Umeclidinium bromide (UMEC); Closed triple therapy; Placebo; Open triple therapy; fluticasone furoate/vilanterol (FF/VI)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF/UMEC/VI closed triple therapy plus Placebo (Experimental): Subjects will receive FF/UMEC/VI, 100 mcg/62.5 mcg/25 mcg and placebo inhalation powder via the dry powder inhaler (DPI), once daily in the morning. Subjects will also receive albuterol/salbutamol as a rescue medication when needed during the treatment period.
  Interventions: Drug: FF/UMEC/VI; Drug: Placebo; Drug: Albuterol/salbutamol
- FF/VI plus UMEC open triple therapy (Active Comparator): Subjects will receive FF/VI, 100 mcg/25 mcg and UMEC, 62.5 mcg inhalation powder via the DPI, once daily in the morning. Subjects will also receive albuterol/salbutamol as a rescue medication when needed during the treatment period.
  Interventions: Drug: FF/VI; Drug: UMEC; Drug: Albuterol/salbutamol

INTERVENTIONS:
Drug: FF/UMEC/VI — This intervention is provided in two strips. First strip contains FF blended with lactose. It is available as dry white powder, 100 mcg per blister. Second strip contains UMEC and VI blended with lactose and magnesium stearate. It is available as dry white powder, 62.5 mcg per blister UMEC, 25 mcg per blister VI. The intervention is inhaled via the DPI, once daily in the morning. DPI contains 30 doses (2 strips with 30 blisters per strip).
  Arms: FF/UMEC/VI closed triple therapy plus Placebo
Drug: FF/VI — This intervention is provided in two strips. First strip contains FF blended with lactose. It is available as dry white powder, 100 mcg per blister. Second strip contains VI blended with lactose and magnesium stearate. It is available as dry white powder, 25 mcg per blister. The intervention is inhaled via the DPI, once daily in the morning. DPI contains 30 doses (2 strips with 30 blisters per strip).
  Arms: FF/VI plus UMEC open triple therapy
Drug: UMEC — This intervention is available in one strip. The strip contains UMEC blended with lactose and magnesium stearate. The formulation is available as dry white powder, 62.5 mcg per blister. The intervention is inhaled via the DPI, once daily in the morning. DPI contains 30 doses (1 strip with 30 blisters).
  Arms: FF/VI plus UMEC open triple therapy
Drug: Placebo — This intervention is available in one strip. The strip contains lactose. The formulation is available as dry white powder. The intervention is inhaled via the DPI, once daily in the morning. DPI contains 30 doses (1 strip with 30 blisters).
  Arms: FF/UMEC/VI closed triple therapy plus Placebo
Drug: Albuterol/salbutamol — This is a rescue medication administered via metered-dose inhaler (MDI) with a spacer which will be used when needed during the study.

SUMMARY:
This multicenter study will be conducted to compare the effect of FF/UMEC/VI with FF/VI plus UMEC on lung function after 24 weeks of treatment. This is a phase IIIB, 24-week, randomized, double-blind, parallel group multicenter study. This study will test the hypothesis that the difference in trough forced expiratory volume in one second (FEV1) between treatment groups is less than or equal to a pre-specified non-inferiority margin. Alternatively, this study will also test the hypothesis that the difference between treatment groups is greater than the margin. The triple therapy of FF/UMEC/VI in a single inhaler is being developed with the aim of providing a new treatment option for the management of advanced Global Initiative for Chronic Obstructive Lung Disease (GOLD) Group D COPD which will reduce the exacerbation frequency, allow for a reduced burden of polypharmacy, convenience, and improve lung function, health related quality of life (HRQoL) and symptom control over established dual/monotherapies. This study has a 2 week run in period where subjects will continue to have their existing COPD medications. At randomization, subjects will discontinue all existing COPD medications and will be assigned to treatment of FF/UMEC/VI, 100 microgram (mcg)/62.5 mcg/25 mcg and placebo or FF/VI, 100 mcg/25 mcg and UMEC, 62.5 mcg in a 1:1 ratio for 24 weeks. Subjects will have clinical visits at Pre-Screening (Visit 0), Screening (Visit 1), Randomization (Week 0, Visit 2), Week 4 (Visit 3), Week 12 (Visit 4) and Week 24 (Visit 5). A follow-up visit will be conducted at 1 week after the end of treatment period or after early withdrawal visit. Approximately, 1020 subjects will be enrolled in this study. There will be two pharmacokinetic (PK) groups (subset A and subset B). Approximately 120 subjects will be assigned to subset A and approximately 60 subjects will be assigned to subset B. The total duration of subject participation will be approximately 27 weeks, consisting of a 2-week run-in period, 24-week treatment period and a 1-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent: A signed and dated written informed consent prior to study participation.

* Type of subject: Outsubject.
* Age: Subjects 40 years of age or older at Screening (Visit 1).
* Gender: Male or female subjects. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as:

* Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy.
* Postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study treatmentand until after the last dose of study treatmentand completion of the follow-up visit.

* COPD Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at Screening (Visit 1) [number of pack years = (number of cigarettes per day divided by 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Screening (Visit 1). Note: Pipe and/or cigar use cannot be used to calculate pack-year history.
* Severity of COPD symptoms: A score of >=10 on the COPD Assessment Test (CAT) at Screening (Visit1).
* Severity of COPD Disease: A post-albuterol/salbutamol FEV1/FVC ratio of <0.70 at Screening (Visit 1).
* Existing COPD maintenance treatment: Subject must be receiving daily maintenance treatment for their COPD for at least 3 months prior to Screening (Visit 1). Note: Subjects receiving only as needed COPD medications are not eligible.
* History of Exacerbations: Subjects must demonstrate: a post-bronchodilator FEV1 <50 percent predicted normal at Screening (Visit 1) and a documented history of >=1 moderate or severe COPD exacerbation in the 12 months prior to Screening or a post-bronchodilator 50 percent =< FEV1 <80 percent predicted normal at Screening (Visit 1) and a documented history of >=2 moderate exacerbations or a documented history of >=1 severe COPD exacerbation (hospitalised) in the 12 months prior to Screening (Visit 1). Notes: Percent predicted will be calculated using the European Respiratory Society Global Lung Function Initiative reference equations; A documented history of a COPD exacerbation (e.g., medical record verification) is a medical record of worsening COPD symptoms that required systemic/oral corticosteroids and/or antibiotics (for a moderate exacerbation) or hospitalisation (for a severe exacerbation). Prior use of antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD, such as increased dyspnoea, sputum volume, or sputum purulence (colour). Subject verbal reports are not acceptable.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD, which is the primary cause of their respiratory symptoms).
* Alpha 1-antitrypsin deficiency: Subjects with alpha1-antitrypsin deficiency as the underlying cause of COPD.
* Other respiratory disorders: Subjects with active tuberculosis are excluded. Subjects with other respiratory disorders (e.g. clinically significant: bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases) are excluded if these conditions are the primary cause of their respiratory symptoms.
* Lung resection: Subjects with lung volume reduction surgery (including procedures such as endobronchial valves) within the 12 months prior to Screening (Visit 1).
* Risk Factors for Pneumonia: immune suppression (e.g. advanced human immune deficiency virus (HIV) with high viral load and low cluster of differentiation 4 (CD4) count, Lupus on immunosuppressants that would increase risk of pneumonia) or other risk factors for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis). Notes: Subjects at a high risk for pneumonia (e.g. very low body mass index (BMI), severely malnourished or very low FEV1) will only be included at the discretion of the investigator.
* Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening (Visit 1) and at least 30 days following the last dose of oral/systemic corticosteroids (if applicable).
* Other Respiratory tract infections that have not resolved at least 7 days prior to Screening (Visit 1).
* Abnormal Chest x-ray: Chest x-ray reveals evidence of pneumonia or a clinically significant abnormality not believed to be due to the presence of COPD, or another condition that would hinder the ability to detect an infiltrate on chest x-ray (e.g. significant cardiomegaly, pleural effusion or scarring). All subjects will have a chest x-ray at Screening (Visit 1) [or historical radiograph or computerised tomography (CT) scan obtained within 3 months prior to Screening (Visit 1). Notes: Subjects who have experienced pneumonia and/or moderate or severe COPD exacerbation within 3 months of Screening (Visit 1) must provide a post pneumonia/exacerbation chest x-ray or have a chest x-ray conducted at Screening (Visit 1); For sites in Germany: If a chest x-ray (or CT scan) within 3 months prior to Screening (Visit 1) is not available, approval to conduct a diagnostic chest x-ray will need to be obtained from the Federal Office for Radiation Protection (BFS).
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Unstable liver disease: ALT >2 times upper limit of normal (ULN); and bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent). Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment). Notes: Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice, or cirrhosis; Chronic stable hepatitis B and C (e.g., presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment) are acceptable if subject otherwise meets entry criteria.
* Unstable or life threatening cardiac disease: subjects with any of the following at Screening (Visit 1) would be excluded: Myocardial infarction or unstable angina in the last 6 months; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class 4 Heart failure.
* Abnormal and clinically significant 12-Lead ECG finding: Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. The investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding that would preclude a subject from entering the trial is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following: atrial fibrillation (AF) with rapid ventricular rate >120 beats per minute (BPM); sustained or nonsustained ventricular tachycardia (VT); Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted).
* Contraindications: A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the investigator contraindicates study participation.
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 3 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 3 year waiting period if the subject has been considered cured by treatment.
* Oxygen therapy: Use of long-term oxygen therapy (LTOT) described as resting oxygen therapy >3 Liters per minute (Oxygen use <= 3 Liters/minute flow is not exclusionary.)
* Medication prior to spirometry: Subjects who are medically unable to withhold their albuterol/salbutamol for the 4-hour period required prior to spirometry testing at each study visit.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Affiliation with investigator site: Study investigators, sub-investigators, and study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete study related materials.
* Medication prior to Screening: Use of the following medications within 30 days prior to Screening (Visit 1) or requirement for their use during the study: Use of long term continuous antibiotic therapy; systemic, oral, parenteral corticosteroids (Intra-spinal and intra-articular injections are allowed); use of any other investigational drug: within 30 days or 5 half lives whichever is longer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1055 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (99):
- Argentina (5):
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (8):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Woodville South, South Australia
  - GSK Investigational Site, Footscray, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
  - GSK Investigational Site, Golden Beach
- France (6):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Pringy
  - GSK Investigational Site, Toulouse
- Germany (16):
  - GSK Investigational Site, Dillingen an der Donau, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Peine, Lower Saxony
  - GSK Investigational Site, Wardenburg, Lower Saxony
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Rheine, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Leipzg, Saxony
- Italy (6):
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, San Sisto (PG), Umbria
- Japan (19):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Mexico (6):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Ciudad de México, State of Mexico
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, México DF
- Poland (6):
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Ostrow Wilekopolski
  - GSK Investigational Site, Tarnów
- Romania (6):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Târgu Mureş
  - GSK Investigational Site, Timișoara
- Russia (12):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petesburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ufa
- South Korea (3):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
  - GSK Investigational Site, Wonju, Gangwon-do,
- Spain (6):
  - GSK Investigational Site, Laredo, Cantabria
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Bremner PR, Birk R, Brealey N, Ismaila AS, Zhu CQ, Lipson DA. Single-inhaler fluticasone furoate/umeclidinium/vilanterol versus fluticasone furoate/vilanterol plus umeclidinium using two inhalers for chronic obstructive pulmonary disease: a randomized non-inferiority study. Respir Res. 2018 Jan 25;19(1):19. doi: 10.1186/s12931-018-0724-0. PMID 29370819
- [Derived] Mehta R, Farrell C, Hayes S, Birk R, Okour M, Lipson DA. Population Pharmacokinetic Analysis of Fluticasone Furoate/Umeclidinium Bromide/Vilanterol in Patients with Chronic Obstructive Pulmonary Disease. Clin Pharmacokinet. 2020 Jan;59(1):67-79. doi: 10.1007/s40262-019-00794-w. PMID 31321713
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 24-week, randomized, double-blind, parallel group multicenter study to compare closed triple therapy Fluticasone Furoate/ Umeclidinium/ Vilanterol Trifenatate (FF/UMEC/VI) with open triple therapy (FF/VI + UMEC), in participants with chronic obstructive pulmonary disease (COPD). This study was conducted across 12 countries.
Pre-assignment Details: A total of 1311 participants were pre-screened, of which 1278 participants were screened (33 pre-screen failures). There were 175 screen failures and 48 Run-in failures. A total of 1055 participants were randomized and received the study treatment.
Groups:
- FF/UMEC/VI 100/62.5/25: Participants received FF/UMEC/VI, 100 micrograms (mcg)/62.5 mcg/25 mcg via ELLIPTA dry powder inhaler (DPI) once daily in morning and placebo inhalation powder via ELLIPTA DPI, once daily in the morning. Participants also received albuterol/salbutamol as a rescue medication when needed during the treatment period.
- FF/VI 100/25 + UMEC 62.5: Participants received FF/VI, 100 mcg/25 mcg via ELLIPTA DPI once daily in morning and UMEC 62.5 mcg inhalation powder via ELLIPTA DPI, once daily in the morning. Participants also received albuterol/salbutamol as a rescue medication when needed during the treatment period.
Period: Overall Study
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 + UMEC 62.5
Started | 527 | 528
Completed | 497 | 496
Not Completed | 30 | 32
Not completed — Adverse Event | 21 | 11
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 6 | 17

BASELINE CHARACTERISTICS:
Groups:
- FF/UMEC/VI 100/62.5/25: Participants received FF/UMEC/VI, 100 mcg/62.5 mcg/25 mcg via ELLIPTA DPI once daily in morning and placebo inhalation powder via ELLIPTA DPI, once daily in the morning. Participants also received albuterol/salbutamol as a rescue medication when needed during the treatment period.
- Total: Total of all reporting groups
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 + UMEC 62.5 | Total
Number analyzed (Participants) | 527 | 528 | 1055
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (8.46) | 65.9 (8.77) | 66.3 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 134 | 270
  Male | 391 | 394 | 785
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 14 | 32
  Asian - East Asian Heritage | 29 | 30 | 59
  Asian - Japanese Heritage | 41 | 38 | 79
  Asian - South East Asian Heritage | 2 | 0 | 2
  White - Arabic/North African Heritage | 1 | 4 | 5
  White - White/Caucasian/European Heritage | 416 | 416 | 832
  American Indian/Alaska Native and Asian and White | 0 | 1 | 1
  American Indian or Alaska Native and White | 20 | 25 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. It was measured using centralized spirometry. FEV1 values at Week 0, pre-dose were considered as Baseline values. Change from Baseline was calculated by subtracting Baseline value from the value at indicated time point. Modified Per Protocol (mPP) Population was used which comprised of all participants in the Intent-to-Treat (ITT) Population, who do not have a full protocol deviation considered to impact efficacy. Data following a moderate/severe COPD exacerbation or pneumonia was excluded from analysis due to the potential impact of the exacerbation or the medications used to treat it. Participants with partial protocol deviations considered to impact efficacy were included in the mPP Population but had their data excluded from analysis from the time of deviation onwards. Analysis was performed using a mixed model repeated measures (MMRM) method.
Time Frame: Baseline and Week 24
Population: mPP Population
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 + UMEC 62.5
Number analyzed (Participants) | 307 | 287
Liter | 0.113 (0.0112) | 0.095 (0.0116)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 vs FF/VI 100/25 + UMEC 62.5; Test type: Non-Inferiority — If the lower bound of the two-sided 95% confidence interval around the (FF/UMEC/VI versus FF/VI+UMEC) treatment difference is above -50 milliliter (mL) then FF/UMEC/VI was to be considered non-inferior to FF/VI+UMEC; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.013 to 0.050], Standard Error of Mean 0.0161 — MMRM method included covariates of Baseline FEV1, stratum (number of long-acting bronchodilators per day during the run-in: 0/1 or 2), visit, geographical region, treatment, visit by treatment and visit by Baseline interaction

2. Secondary Outcome: Percentage of Responders Based on the Saint (St) George Respiratory Questionnaire (SGRQ) Total Score at Week 24
Description: SGRQ is a disease-specific questionnaire designed to measure impact of respiratory disease and its treatment on health related quality of life (HRQoL) of participants with COPD. It contains 14 questions with a total of 40 items grouped into domains (Symptoms, Activity and Impacts). SGRQ total score was calculated as 100 multiplied by summed weights from all positive items divided by sum of weights for all items in questionnaire. It ranges from 0 to 100, higher score indicates poor HRQoL. Response was defined as an SGRQ total score of >=4 units below Baseline. Non response was defined as a SGRQ total score <4 units below Baseline or a missing SGRQ total score with no subsequent on treatment scores. ITT Population comprised of randomized participants, excluding those who were randomized in error. A participant screened or run-in failure and also randomized was considered to be randomized in error. Analysis was performed using a generalized linear mixed model with a logit link function.
Time Frame: Week 24
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 + UMEC 62.5
Number analyzed (Participants) | 489 | 483
Percentage of Participants | 50 | 51
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 vs FF/VI 100/25 + UMEC 62.5; Test type: Other; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.71 to 1.20] — Analysis included covariates of treatment group, stratum (number of long-acting bronchodilators per day during the run-in: 0/1 or 2), geographical region, visit, Baseline, Baseline by visit and treatment by visit interactions

3. Secondary Outcome: Change From Baseline in SGRQ Total Score at Week 24
Description: SGRQ is a disease-specific questionnaire designed to measure impact of respiratory disease and its treatment on HRQoL of participants with COPD. It contains 14 questions with a total of 40 items grouped into domains (Symptoms, Activity and Impacts). SGRQ total score was calculated as 100 multiplied by summed weights from all positive items divided by sum of weights for all items in questionnaire. It ranges from 0 to 100, higher score indicates poor HRQoL. Values at Week 0, pre-dose were considered as Baseline values. Change from Baseline was calculated by subtracting Baseline value from the value at indicated time point. Analysis was performed using a MMRM method including covariates of Baseline SGRQ Total score, stratum (number of long-acting bronchodilators per day during the run-in: 0/1 or 2), visit, geographical region, treatment, visit by treatment and visit by Baseline interaction.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 + UMEC 62.5
Number analyzed (Participants) | 489 | 483
Scores on a scale | -5.841 (0.5870) | -4.935 (0.5904)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 vs FF/VI 100/25 + UMEC 62.5; Test type: Other; Least Square Mean Difference = -0.906, 95% CI 2-sided [-2.540 to 0.728], Standard Error of Mean 0.8327 — Analysis performed using a repeated measures model with covariates of Baseline SGRQ, stratum (number of long-acting bronchodilators per day during the run-in: 0/1 or 2), visit, geographical region, treatment, visit by treatment and visit by Baseline

4. Secondary Outcome: Percentage of Responders Based on Transitional Dyspnea Index (TDI) Focal Score at Week 24
Description: The TDI measures changes in the participant's dyspnea. TDI focal score was calculated as the sum of the ratings recorded for each of the 3 individual scales (Functional Impairment, Magnitude of Task, Magnitude of Effort). Each of these scales had a possible score ranging from -6 to +6. lower scores indicating more impairment. TDI focal score was calculated as the sum of the 3 individual scores and then divided by 2 (so the range of the TDI focal score is -9 to +9). The lower the score, the more deterioration in severity of dyspnea. If a score is missing for any of the three scales, then the TDI focal score was set to missing. A participant was considered as a responder if the on-treatment TDI focal score was at least 1 unit at that visit. Non-response was defined as a TDI focal score of less than 1 unit or a missing TDI focal score with no subsequent non-missing on-treatment scores. Analysis was performed using a generalized linear mixed model with a logit link function.
Time Frame: Week 24
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 + UMEC 62.5
Number analyzed (Participants) | 482 | 481
Percentage of Participants | 56 | 56
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 vs FF/VI 100/25 + UMEC 62.5; Test type: Other; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.72 to 1.25] — Include covariates of treatment group, stratum (number of long-acting bronchodilators/ day during the run-in: 0/1 or 2), geographical region, visit, Baseline dyspnea index (BDI) focal score, BDI focal score/ visit and treatment/ visit interactions

5. Secondary Outcome: TDI Focal Score at Week 24
Description: The TDI measures changes in the participant's dyspnoea. TDI focal score was calculated as the sum of the ratings recorded for each of the 3 individual scales (Functional Impairment, Magnitude of Task, Magnitude of Effort). Each of these scales had a possible score ranging from -6 to +6. lower scores indicating more impairment. TDI focal score was calculated as the sum of the 3 individual scores and then divided by 2 (so the range of the TDI focal score is -9 to +9). The lower the score, the more deterioration in severity of dyspnea. If a score is missing for any of the three scales, then the TDI focal score was set to missing. Analysis was performed using a repeated measures model.
Time Frame: Week 24
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 + UMEC 62.5
Number analyzed (Participants) | 482 | 481
Scores on a scale | 2.029 (0.1252) | 1.892 (0.1254)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 vs FF/VI 100/25 + UMEC 62.5; Test type: Other; Mean Difference (Final Values) = 0.137, 95% CI 2-sided [-0.211 to 0.485], Standard Error of Mean 0.1773 — Analysis included covariates of BDI focal score, stratum (number of long-acting bronchodilators per day during the run-in: 0/1 or 2), visit, geographical region, treatment, visit by treatment and visit by BDI Focal score interactions

6. Secondary Outcome: Time to First Moderate or Severe Exacerbation
Description: COPD exacerbations were identified based on the investigator's clinical judgment. Worsening symptoms of COPD that required treatment with oral/systemic corticosteroids and/or antibiotics were considered as moderate exacerbation. Worsening symptoms of COPD that required treatment with in-subject hospitalization was considered as severe exacerbation. Hazard ratio and 95% confidence interval (CI) is from a Cox proportional hazards model with covariates of treatment group, sex, exacerbation history (0, 1, >=2 moderate/severe exacerbations, prior year), smoking status (screening), stratum (number of long-acting bronchodilators per day during the run-in: 0/1 or 2), geographical region and percent predicted FEV1 at Baseline. Median and inter-quartile range (first and third quartile) have been presented.
Time Frame: Up to 25 weeks
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 + UMEC 62.5
Number analyzed (Participants) | 527 | 528
Days | NA [166 to NA] — As <50% of participants experienced the event within a treatment, median and third-quartile of time to first moderate or severe exacerbation are displayed as NA (not applicable) for that treatment. | NA [150 to NA] — As <50% of participants experienced the event within a treatment, median and third-quartile of time to first moderate or severe exacerbation are displayed as NA (not applicable) for that treatment.
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 vs FF/VI 100/25 + UMEC 62.5; Test type: Other; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.68 to 1.12] — Analysis was performed using a Cox proportional hazards model

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs (nSAEs) were collected from start of study treatment (Week 0) until Week 25 including 1 Week of follow-up.
Description: On-treatment SAEs and nSAEs were reported for ITT Population.
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 + UMEC 62.5
All-Cause Mortality (participants affected / at risk) | 7/527 | 5/528
Serious Adverse Events (participants affected / at risk) | 55/527 | 60/528
Other Adverse Events (participants affected / at risk) | 122/527 | 125/528
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/UMEC/VI 100/62.5/25 (N=527) | FF/VI 100/25 + UMEC 62.5 (N=528)
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Degenerative aortic valve disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Gastritis hypertrophic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 | 2
Influenza (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 9 | 13
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Superinfection (Infections and infestations) | 0 | 1
Toxic shock syndrome (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
X-ray abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Organic brain syndrome (Psychiatric disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 24 | 32
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aortic aneurysm (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/UMEC/VI 100/62.5/25 (N=527) | FF/VI 100/25 + UMEC 62.5 (N=528)
Viral upper respiratory tract infection (Infections and infestations) | 56 | 52
Upper respiratory tract infection (Infections and infestations) | 18 | 24
Influenza (Infections and infestations) | 16 | 17
Pharyngitis (Infections and infestations) | 12 | 16
Headache (Nervous system disorders) | 32 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02729051/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT02729051/SAP_001.pdf